CLINICAL TRIAL: NCT04833166
Title: A Randomized Controlled Trial Comparing Full Glottis View vs. Partial Glottis View During Intubation Using CMAC D-Blade Video Laryngoscope in Simulated Cervical Injury Patient
Brief Title: Comparing Full vs. Partial Glottis View Using CMAC D-Blade Video Laryngoscope in Simulated Cervical Injury Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr. Cheong Chao Chia, Doctor/ Clinical Anaesthesiologist/ Clinical Lecturer, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MREC: 202093-9041
Record Dates: First submitted 2021-03-01; First posted 2021-04-06 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Intubation; Difficult or Failed; Airway Complication of Anesthesia
Keywords: Glottic view; Intubation time; C MAC D- blade

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full glottic view on CMAC- D blade (Experimental): Deliberately obtaining a full glottis view is deﬁned as negotiation and advancement of CMAC D blade tip positioned at the vallecula. Occasionally, external laryngeal pressure may be needed to assist in obtaining a full glottic view. The full glottic view is defined as a percentage of glottic opening (POGO) approximate 100%.
  Interventions: Device: CMAC D-blade videolaryngoscope with full or partial glottic view
- Partial glottic view on CMAC- D blade (Active Comparator): The partial glottis view is deﬁned as a percentage of glottic opening <50%. This is achieved by deliberately position the CMAC D-blade tip proximally away from the vallecular.
  Interventions: Device: CMAC D-blade videolaryngoscope with full or partial glottic view

INTERVENTIONS:
Device: CMAC D-blade videolaryngoscope with full or partial glottic view — Deliberate achieving full or partial glottic view on C MAC D-blade video laryngoscope and comparing time and ease of intubation with both arms

SUMMARY:
Direct laryngoscope requires proper alignment of the oro-pharyngeal-laryngeal axis to provide an optimal glottic view for intubation. However, in cervical spine patients, this alignment is not possible thus resulting in an increased risk of fail intubations.

D-blade comes with an elliptically tapered blade shape rising at the distal end to provide better glottic visualization in comparison with direct laryngoscopes. Hence, CMAC D-blade is preferred in simulated cervical spine injury where intubator needs to maintain a neutral neck position. However, intubation time may be significantly longer due to difficulty in negotiating the endotracheal tube pass vocal cord and impingement of endotracheal tube to the anterior wall of trachea.

There is a study published Glidescope which is also a hyperangulated videolaryngoscope suggested that obtaining a partial glottic view of larynx may facilitate a faster and easier tracheal intubation when compare to a full glottis view. The aim of this study is to clinically evaluate the time of tracheal intubation in relation to the full glottic view vs. partial glottic view which is deliberately obtained when using CMAC D-blade video laryngoscopy in simulated cervical spine injury.

DETAILED DESCRIPTION:
Direct laryngoscope requires proper alignment of the oro-pharyngeal-laryngeal axis to provide the best laryngeal view for intubation. In cervical spine patients, this alignment is not possible resulting in an increased risk of failed intubations. Difficult intubation and failed tracheal intubation are among the major causes of morbidity and mortality associated with anesthesia.

In recent years, video laryngoscope has played an increasingly important role in the management of patients with unanticipated difficult or failed endotracheal intubation. When compared with a direct laryngoscope, the video laryngoscope achieved a better view of the glottis and a high rate of successful intubation.

On comparing the C-MAC with the conventional Macintosh blade, a conventional C-MAC Macintosh blade 3 and D-blade have a blade angulation of 18° and 40° in the D-blade respectively. In addition, with D-blade is an elliptically tapered blade-shaped rising to distal.

This highly angulated C-MAC D blade provides a better glottic visualization in comparison to the direct laryngoscopes and in simulated cervical spine injury. This resulted in successful intubation in routine induction of anesthesia and rescue intubation in patients with difficult airway with C-MAC D Blade. But in terms of intubation time, study has shown a significantly shorter time with C-MAC D Blade compared with other indirect laryngoscopes. This may be due to a common problem seen in indirect video laryngoscopy whereby a good glottic view does not always allow advancing the tube into the trachea.

A study has been conducted on Glidescope which is also a hyperangulated blade suggested that obtaining a partial glottic view of larynx may facilitate a faster and easier tracheal intubation when compare to a full glottis view. Randomised controlled trial also showed that GlideScope and C-MAC D blade video laryngoscope using manual inline axial stabilization (MIAS) for tracheal intubation in patients with cervical spine injury/pathology were equally efficacious.

The aim of this study is to clinically evaluate the time of tracheal intubation in relation to deliberately obtained full glottic view vs. partial glottic view when using CMAC D-blade video laryngoscopy in simulated cervical spine injury.

ELIGIBILITY:
Inclusion Criteria:

* All patients with American Society of Anaesthesiologist (ASA) physical status I-III
* Age (≥21-75 years old)
* General anaesthesia requiring tracheal intubation
* Provide written consent to participate in the study

Exclusion Criteria:

* Pregnancy
* Body mass index (BMI) ≥ 35
* Condition requires rapid sequence induction
* Need for fibreoptic intubation
* Need for nasal intubation
* Documented difficult airway during previous surgery
* Recent (3 months) active ischemic heart disease
* Recent (3 months) cerebrovascular disease
* Acute exacerbation of respiratory disease (eg. Uncontrolled asthma, Chronic Obstructive Pulmonary Disease)

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Intubation time | during the intervention
  This is the time taken from CMAC laryngoscope blade passes patient's lip until the recording of first end tidal CO2 (EtCO2); assessed up to 120 seconds.
First attempt successful intubation attempt | during the intervention
  First intubation attempt success rate between two groups; assessed up to maximum 2 attempts

SECONDARY OUTCOMES:
Time to obtain glottic view | during the intervention
  Time taken for from CMAC laryngoscope blade passes patient's lip until achieving assigned laryngoscopic view; assessed up to 120 seconds
Hemodynamic changes | immediately after the intervention
  Blood pressure, mean arterial pressure and heart rate recorded 1 min, 2.5 min then 5 min post intubation
Airway trauma | immediately after the surgery
  Incidence of oral mucosal trauma, lip laceration, dental laceration; assessed up to discharge from operating theatre.

CONTACTS AND LOCATIONS:
Overall Officials: Siu Min Lim, MMed Master, Study Director — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adnet F, Borron SW, Lapostolle F, Lapandry C. The three axis alignment theory and the "sniffing position": perpetuation of an anatomic myth? Anesthesiology. 1999 Dec;91(6):1964-5. doi: 10.1097/00000542-199912000-00060. No abstract available. PMID 10598648
- [Background] Criswell JC, Parr MJ, Nolan JP. Emergency airway management in patients with cervical spine injuries. Anaesthesia. 1994 Oct;49(10):900-3. doi: 10.1111/j.1365-2044.1994.tb04271.x. PMID 7802192
- [Background] Caplan RA, Posner KL, Ward RJ, Cheney FW. Adverse respiratory events in anesthesia: a closed claims analysis. Anesthesiology. 1990 May;72(5):828-33. doi: 10.1097/00000542-199005000-00010. PMID 2339799
- [Background] Mort TC. Emergency tracheal intubation: complications associated with repeated laryngoscopic attempts. Anesth Analg. 2004 Aug;99(2):607-13, table of contents. doi: 10.1213/01.ANE.0000122825.04923.15. PMID 15271750
- [Background] Stroumpoulis K, Pagoulatou A, Violari M, Ikonomou I, Kalantzi N, Kastrinaki K, Xanthos T, Michaloliakou C. Videolaryngoscopy in the management of the difficult airway: a comparison with the Macintosh blade. Eur J Anaesthesiol. 2009 Mar;26(3):218-22. doi: 10.1097/EJA.0b013e32831c84d1. PMID 19237983
- [Background] Su YC, Chen CC, Lee YK, Lee JY, Lin KJ. Comparison of video laryngoscopes with direct laryngoscopy for tracheal intubation: a meta-analysis of randomised trials. Eur J Anaesthesiol. 2011 Nov;28(11):788-95. doi: 10.1097/EJA.0b013e32834a34f3. PMID 21897263
- [Background] Lewis SR, Butler AR, Parker J, Cook TM, Schofield-Robinson OJ, Smith AF. Videolaryngoscopy versus direct laryngoscopy for adult patients requiring tracheal intubation: a Cochrane Systematic Review. Br J Anaesth. 2017 Sep 1;119(3):369-383. doi: 10.1093/bja/aex228. PMID 28969318
- [Background] Cavus E, Neumann T, Doerges V, Moeller T, Scharf E, Wagner K, Bein B, Serocki G. First clinical evaluation of the C-MAC D-Blade videolaryngoscope during routine and difficult intubation. Anesth Analg. 2011 Feb;112(2):382-5. doi: 10.1213/ANE.0b013e31820553fb. Epub 2010 Dec 14. PMID 21156978
- [Background] Jain D, Dhankar M, Wig J, Jain A. Comparison of the conventional CMAC and the D-blade CMAC with the direct laryngoscopes in simulated cervical spine injury--a manikin study. Braz J Anesthesiol. 2014 Jul-Aug;64(4):269-74. doi: 10.1016/j.bjane.2013.06.005. Epub 2013 Dec 25. PMID 24998112
- [Background] Serocki G, Neumann T, Scharf E, Dorges V, Cavus E. Indirect videolaryngoscopy with C-MAC D-Blade and GlideScope: a randomized, controlled comparison in patients with suspected difficult airways. Minerva Anestesiol. 2013 Feb;79(2):121-9. Epub 2012 Oct 2. PMID 23032922
- [Background] van Zundert A, Maassen R, Lee R, Willems R, Timmerman M, Siemonsma M, Buise M, Wiepking M. A Macintosh laryngoscope blade for videolaryngoscopy reduces stylet use in patients with normal airways. Anesth Analg. 2009 Sep;109(3):825-31. doi: 10.1213/ane.0b013e3181ae39db. PMID 19690253
- [Background] Gu Y, Robert J, Kovacs G, Milne AD, Morris I, Hung O, MacQuarrie K, Mackinnon S, Adam Law J. A deliberately restricted laryngeal view with the GlideScope(R) video laryngoscope is associated with faster and easier tracheal intubation when compared with a full glottic view: a randomized clinical trial. Can J Anaesth. 2016 Aug;63(8):928-37. doi: 10.1007/s12630-016-0654-6. Epub 2016 Apr 18. PMID 27090535
- [Derived] Cheong CC, Ong SY, Lim SM, Wan A WZ, Mansor M, Chaw SH. Partial vs full glottic view with CMACTM D blade intubation of airway with simulated cervical spine injury: a randomized controlled trial. Expert Rev Med Devices. 2023 Feb;20(2):151-160. doi: 10.1080/17434440.2023.2174850. Epub 2023 Feb 6. PMID 36715659